CLINICAL TRIAL: NCT05167019
Title: Coaching Doctors to Improve Ethical Decision-making in Adult Hospitalized Patients Potentially Receiving Excessive Treatment: a Step Wedge Cluster Randomized Trial in 10 Departments of the Ghent University Hospital (CODE)
Brief Title: Coaching Doctors in Ethical Decision-making (CODE)
Acronym: CODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: BC-09828
Record Dates: First submitted 2021-10-01; First posted 2021-12-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: End of Life; Interdisciplinary Communication; Leadership
Keywords: Treatment limitation decisions; Interdisciplinary collaboration; Coaching; Self-reflective and empowering leadership; Ethical climate; Prognostic uncertainty
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Sample size for this stepped wedge randomised controlled trial is listed for patients potentially receiving excessive treatment (n=1700) together with one of their relatives who will be identified by junior doctors (n=75) , senior doctors (n=75) and nurses (n= 600) working in 10 departments of the Ghent university hospital during a 12 months period. Junior and senior doctors working in each department will be coached in self-reflective and empowering leadership, and in managing group dynamics with regard to patients potentially receiving excessive treatment for whom they are in charge of during a 4 month period. The impact of the intervention on the quality of ethical decision-making will be assessed at the patient (n=1700), relatives (n=1700) and team level (n=750).
Who Masked: Participant
Masking Description: Patients will be blinded to the 4 months intervention period in junior and senior doctors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care
  Interventions: Other: Usual care
- The CODE intervention (Experimental): The CODE intervention consists of 4 items, of which individual coaching sessions of 1 hour. In total each doctor taking care of hospitalized patients will be able to receive maximum 16 individual coaching sessions during the 4 months intervention period (one weekly). Every doctor will be invited to participate to at least 8 coaching sessions, to be extended on request, during the intervention period.
  Interventions: Behavioral: CODE intervention

INTERVENTIONS:
Behavioral: CODE intervention — The CODE intervention consists of 1) One interactive session of 2 to 3 hrs focusing on the concepts of medical-ethical decision-making, the psychological challenge of dealing with ethically sensitive medical topics, and empowering leadership. 2) Observation and debrief of the interdisciplinary meeting to enhance self-reflection on empowering leadership and managing group dynamics. 3) Individual coaching on the spot in self-reflective and empowering leadership and in managing groups dynamics with regard to ethical decision-making about patients who are perceived to receive excessive treatment during the intervention period, and in absence of such patients, every item with regard to ethical decision-making that is important for the coachee. 4) During the intervention coaches and doctors in charge will be informed of the presence of a patient potentially receiving excessive treatment in their ward by an electronic alert.
  Arms: The CODE intervention
Other: Usual care — The control group will receive usual care in which the quality of the ethical decision-making is determined by the clinical team according to their usual practice. Except from a treatment-limitation-decisions guideline which focuses on the legal and deontological framework, no other guideline with regard to ethical decision-making has been implemented at the Ghent University Hospital. In one ward (geriatrics), there is a ongoing project in which a clinical nurse specialist stimulates and performes advance care planning conversations with patient and/or relatives at request of the team and who organizes debriefings when needed based on the ethical concerns of the nurses.
  Arms: Usual care

SUMMARY:
Over the last few decades the fast technical and medical progress poses a significant challenge to doctors, who are asked to find the right balance between life-prolonging and palliative care. Previous studies suggest that doctors (unconsciously) prefer to remain prognostically uncertain rather than to gather the information that is required to reduce uncertainty and to effectively timely take decisions in the team for the benefit of the patient. To obtain all that information, the doctor in charge of the patient needs to empower clinicians to speak up while guarantying a safe environment. However, creating a safe climate which enhances inter-professional shared decision-making for the benefit of the patient requires specific self-reflective and empowering leadership skills (including the management of group dynamics in the interdisciplinary team).

The aim of this study is to investigate whether coaching doctors in self-reflective and empowering leadership, and in the management of team dynamics with regard to adult hospitalized patients potentially receiving excessive treatment during 4 months 1) improves ethical decision-making (primary objective) and 2) reduces the burden on patients, relatives, clinicians and the society (secondary objective). The improvement in quality of ethical decision-making will be assessed objectively via the incidence of written do-not-intubate and -resuscitate orders (first primary endpoint) in patients potentially receiving excessive treatment and subjectively via the ethical decision-making climate questionnaire that will be filled out by the team (second primary endpoint). In line with the DISPROPRICUS study, patients potentially receiving excessive treatment will be defined as patients who are perceived as receiving excessive treatment by two or more different clinicians in charge of the patient. The probability of being alive, at home with a good quality of life one year after admission was only 7% in patients potentially receiving excessive treatment in this study. Therefore, perceptions of excessive treatment by two or more clinicians are used in this study as a signal to initiate (self-)reflection in team about the quality of care that is provided to the patient and whether the treatment is in balance with the medical condition of the patient and the patient's goal of care

.

ELIGIBILITY:
Inclusion criteria

1. Clinicians' level : doctors (including department head) and nurses (including head nurses) taking care of adult hospitalized patients in the 10 participating departments
2. Patients' level : first hospitalization of adult patients who are potentially receiving excessive treatment.
3. Family level : family of adult patients who are potentially receiving excessive treatment

Exclusion criteria :

1. Clinicians'level : no exclusion criteria
2. Patients' level : patients who cannot understand Dutch questionnaires
3. Family : persons who cannot understand Dutch questionnaires

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Incidence of written do-not-intubate and -resuscitate (DNIR) order between hospital admission and the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Ethical decision-making climate questionnaire (EDMCQ) | at the start and end of the 12 month study period
  Clinician specific endpoint. Factorscores on 7 domains, which is normally distributed, centred at mean of zero, with standard deviation 5.5 (minimum score -25, maximum score 25). Higher scores iindicate higher quality of ethical decision-making

SECONDARY OUTCOMES:
Incidence of death one year after first hospital admission | 12 months after first hospital admission
  Patient-specific endpoint
Percentage of patients who achieved the combined one year patient outcome (dead, not at home or utility <0.5 according to the European Quality-of-life 5 dimension instrument (Euro-QOL-5D). | 12 months after first hospital admission
  Patient-specific endpoint
Number of days admitted in the hospital up the end of the first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Pain according to the Numeral rating scale (NRS) : sum of the average daily score up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint. Single-item assessment of pain ranging from 0 (no pain) to 10 (worst possible pain).
Pain according to the Numeral rating scale (NRS) : number of days with an average score > 3 up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint. Single-item assessment of pain ranging from 0 (no pain) to 10 (worst possible pain).
Potentially inappropriate or burdersome treatments : incidence of achieving the combined patient burdersome treatment endpoint (achieving outcome 9,10,11,12,13,14,15 or 16) up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of receiving cardio-pulmonary resuscitation up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of admission in the intensive care unit up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of invasive mechanical ventilation in the intensive care unit up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of non-invasive mechanical ventilation in the intensive care unit up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of receiving dialysis up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of receiving a surgical procedure up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of receiving a chemotherapeutic treatment up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdersome treatments : incidence of receiving a radiotherapeutic treatment up to the end of first hospital stay | at the end of the 12 months study period
  Patient-specific endpoint
Satisfaction according to the European Family Satisfaction in the ICU score (Euro FS) | 3 weeks after hospital discharge
  Patient-specific endpoint. The investigators will use the single-item assessment of satisfaction of this score ranging from 0 to 10. Higher values indicate higher satisfaction
Hospital anxiety and depression scale (HADS) | 3 weeks after hospital discharge
  Patient-specific endpoint. This score is interpreted as follows : 0-7 (normal), 8-10 (mild), 11-21 (moderate to severe)
European quality of dying and death family questionnaire (Euro-QODD nurse) | within 1 week after death
  Patient-specific endpoint filled out by nurses. The investigators will use the single-item assessment of quality of dying and death of this score ranging from 0 to 10. Higher values indicate higher quality
European quality of dying and death family questionnaire (Euro-QODD family) | 3 weeks after the patient's death
  Patient-specific endpoint filled out by the relatives. The investigators will use the single-item assessment of quality of dying and death of this score ranging from 0 to 10. Higher values indicate higher quality
Satisfaction according to the European Family Satisfaction in the ICU score (Euro FS) | 3 weeks after the patient's hospital discharge
  Family-specific endpoint. The investigators will use the single-item assessment of satisfaction of this score ranging from 0 to 10. Higher values indicate higher satisfaction
Hospital anxiety and depression scale (HADS) | 3 weeks after the patient's hospital discharge
  Family-specific endpoint. This score is interpreted as follows : 0-7 (normal), 8-10 (mild), 11-21 (moderate to severe)
Impact of events scale-revised (IES-R) | 3 weeks after the patient's death
  Family-specific endpoint. This score is interpreted as follows: Low risk (0-11), moderate risk (12-32), high risk (33 or higher) for post-traumatic stress disorder.
Percentage of (mild-moderate-severe-extreme) stress related to a perception of excessive treatment | at the end of the 12 month study period
  Clinician-specific endpoint
Percentage of clinicians with intention of leaving their job | at the start and end of the 12 month study period
  Clinician-specific endpoint
Percentage of clinicians with sick leave | at the start and end of the 12 month study period
  Team-specific endpoint
Ethical pratice score | at the start and end of the 12 month study period
  Team-specific endpoint. This scores consist of 12 items. The investigators will use the 10 department specific items (minus the 2 country-specific items). This score ranges from 0 to 10 with higher scores indicating a higher degree of ethical pratice organization
Health-care utilization : total hospital cost by the hospital billing record up to the end of first hospital stay | at the end of the 12 months study period
  Society-specific endpoint
Health-care utilization : total number of emergency department visits | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of hospital admissions | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of admissions in the intensive care unit | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of days in the hospital | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of days in the intensive care unit | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of dialyses | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of surgical procedures | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of chemotherapeutic treatments | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of radiotherapeutic treatments | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of blood analyses | 12 months after first hospital discharge
  Society-specific endpoint
Health-care utilization : total number of radiological investigations | 12 months after first hospital discharge
  Society-specific endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Benoit, MD,PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Background] Smith AK, White DB, Arnold RM. Uncertainty--the other side of prognosis. N Engl J Med. 2013 Jun 27;368(26):2448-50. doi: 10.1056/NEJMp1303295. No abstract available. PMID 23802514
- [Background] Van den Bulcke B, Piers R, Jensen HI, Malmgren J, Metaxa V, Reyners AK, Darmon M, Rusinova K, Talmor D, Meert AP, Cancelliere L, Zubek L, Maia P, Michalsen A, Decruyenaere J, Kompanje EJO, Azoulay E, Meganck R, Van de Sompel A, Vansteelandt S, Vlerick P, Vanheule S, Benoit DD. Ethical decision-making climate in the ICU: theoretical framework and validation of a self-assessment tool. BMJ Qual Saf. 2018 Oct;27(10):781-789. doi: 10.1136/bmjqs-2017-007390. Epub 2018 Feb 23. PMID 29475979
- [Background] Benoit DD, Jensen HI, Malmgren J, Metaxa V, Reyners AK, Darmon M, Rusinova K, Talmor D, Meert AP, Cancelliere L, Zubek L, Maia P, Michalsen A, Vanheule S, Kompanje EJO, Decruyenaere J, Vandenberghe S, Vansteelandt S, Gadeyne B, Van den Bulcke B, Azoulay E, Piers RD; DISPROPRICUS study group of the Ethics Section of the European Society of Intensive Care Medicine. Outcome in patients perceived as receiving excessive care across different ethical climates: a prospective study in 68 intensive care units in Europe and the USA. Intensive Care Med. 2018 Jul;44(7):1039-1049. doi: 10.1007/s00134-018-5231-8. Epub 2018 May 28. PMID 29808345
- [Background] Piers RD, Azoulay E, Ricou B, DeKeyser Ganz F, Max A, Michalsen A, Azevedo Maia P, Owczuk R, Rubulotta F, Meert AP, Reyners AK, Decruyenaere J, Benoit DD; Appropricus Study Group of the Ethics Section of the European Society of Intensive Care Medicine. Inappropriate care in European ICUs: confronting views from nurses and junior and senior physicians. Chest. 2014 Aug;146(2):267-275. doi: 10.1378/chest.14-0256. PMID 24832567
- [Background] Palda VA, Bowman KW, McLean RF, Chapman MG. "Futile" care: do we provide it? Why? A semistructured, Canada-wide survey of intensive care unit doctors and nurses. J Crit Care. 2005 Sep;20(3):207-13. doi: 10.1016/j.jcrc.2005.05.006. PMID 16253788
- [Background] Jensen HI, Hebsgaard S, Hansen TCB, Johnsen RFA, Hartog CS, Soultati I, Szucs O, Wilson ME, van den Bulcke B, Benoit DD, Piers R. Perceptions of Ethical Decision-Making Climate Among Clinicians Working in European and U.S. ICUs: Differences Between Nurses and Physicians. Crit Care Med. 2019 Dec;47(12):1716-1723. doi: 10.1097/CCM.0000000000004017. PMID 31625980
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Jensen HI, Gerritsen RT, Koopmans M, Downey L, Engelberg RA, Curtis JR, Spronk PE, Zijlstra JG, Ording H. Satisfaction with quality of ICU care for patients and families: the euroQ2 project. Crit Care. 2017 Sep 7;21(1):239. doi: 10.1186/s13054-017-1826-7. PMID 28882192
- [Background] Gerritsen RT, Jensen HI, Koopmans M, Curtis JR, Downey L, Hofhuis JGM, Engelberg RA, Spronk PE, Zijlstra JG. Quality of dying and death in the ICU. The euroQ2 project. J Crit Care. 2018 Apr;44:376-382. doi: 10.1016/j.jcrc.2017.12.015. Epub 2017 Dec 26. PMID 29291585
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] van der Ploeg E, Mooren TT, Kleber RJ, van der Velden PG, Brom D. Construct validation of the Dutch version of the impact of event scale. Psychol Assess. 2004 Mar;16(1):16-26. doi: 10.1037/1040-3590.16.1.16. PMID 15023089
- [Derived] Piers R, Dillen L, Goethals K, Lievrouw A, Versluys K, De Pauw A, Jacobs C, Moors I, Offner F, Velghe A, Van Den Noortgate N, Depuydt P, Druwe P, Hemelsoet D, Meurs A, Malotaux J, Van Biesen W, Verbeke F, Derom E, Stevens D, De Pauw M, Tromp F, Van Vlierberghe H, Geboes K, Manesse F, Vanheule S, Benoit DD. Coaching doctors to improve ethical decision-making in adult hospitalized patients potentially receiving excessive treatment: Process evaluation study of the CODE intervention in doctors and nurses working in ten acute hospital wards. PLoS One. 2025 Dec 8;20(12):e0337801. doi: 10.1371/journal.pone.0337801. eCollection 2025. PMID 41359551
- [Derived] Benoit DD, De Pauw A, Jacobs C, Moors I, Offner F, Velghe A, Van Den Noortgate N, Depuydt P, Druwe P, Hemelsoet D, Meurs A, Malotaux J, Van Biesen W, Verbeke F, Derom E, Stevens D, De Pauw M, Tromp F, Van Vlierberghe H, Callebout E, Goethals K, Lievrouw A, Liu L, Manesse F, Vanheule S, Piers R. Coaching doctors to improve ethical decision-making in adult hospitalized patients potentially receiving excessive treatment. The CODE stepped-wedge cluster randomized controlled trial. Intensive Care Med. 2024 Oct;50(10):1635-1646. doi: 10.1007/s00134-024-07588-0. Epub 2024 Sep 4. PMID 39230678